CLINICAL TRIAL: NCT00390910
Title: Study to Assess the Safety and Immunogenicity of GSK Biologicals 10-valent Pneumococcal Conjugate Vaccine When Co-administered With DTPa-HBV-IPV/Hib (Infanrix-Hexa) Vaccine in Preterm Infants as a 3-dose Primary Immunization Course During the First 6 Months of Life.
Brief Title: Study to Evaluate the Safety and Immunogenicity of a 10-valent Pneumococcal Conjugate Vaccine in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107737
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2017-05

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal vaccine; Preterm; Safety; Pneumococcal disease; Immunogenicity
MeSH Terms: conditions — Streptococcal Infections; Premature Birth; Pneumococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (3):
- Synflorix™ + Infanrix™ hexa Group I (Experimental): Very preterm infants born after a gestation period of 27-30 weeks (189-216 days)
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Infanrix hexa
- Synflorix™ + Infanrix™ hexa Group II (Experimental): Mild pretem infants born after a gestation period of 31-36 weeks (217-258 days)
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Infanrix hexa
- Synflorix™ + Infanrix™ hexa Group III (Experimental): Infants born after a gestation period of more than 36 weeks (more than 258 days)
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Infanrix hexa

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A — Intramuscular injection, 3 doses
Biological: Infanrix hexa — Intramuscular injection, 3 doses
  Other Names: DTPa-HBV-IPV/Hib

SUMMARY:
This study aims to evaluate the safety, reactogenicity and immunogenicity of GlaxoSmithKline (GSK) Biologicals´ 10-valent pneumococcal conjugate vaccine when co-administered with diphtheria, tetanus, acellular pertussis-hepatitis B virus-inactivated polio virus/Haemophilus influenzae type b (DTPa-HBV-IPV/Hib) vaccine in preterm infants as a 3-dose primary immunization course during the first 6 months of life.

This protocol posting deals with objectives & outcome measures of the primary study. The objectives & outcome measures of the Booster study are presented in a separate protocol posting (NCT number = 00609492)

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol
* A male or female between, and including, 8-16 weeks (56-118 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Born after a gestation period of >27 weeks (at least 189 days).
* If full term born, healthy subjects as established by medical history and clinical examination before entering into the study
* If premature, medically stable condition (not requiring significant medical support or ongoing management for debilitating disease and having demonstrated a clinical course of sustained recovery).

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccines, or planned use during the study period
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs from birth to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol, during the period starting from one month before the first dose of vaccines and up to Visit 6.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, Neisseria meningitidis and/or Streptococcus pneumoniae with the exception of vaccines where the first dose can be given within the first two weeks of life according to the national recommendations
* History of or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio, Haemophilus influenzae type b disease, Neisseria meningitidis.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurologic disorders or seizures (this criterion does not apply to subjects who have had a single, uncomplicated febrile convulsion in the past).
* Acute disease at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins, with the exception of monoclonal antibodies against RSV, and/or any blood products within one month preceding the first dose of study vaccines or planned administration during the active phase of the study.

Ages: 8 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 286 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2007-07-02 (Actual); Study Completion 2008-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Rio/Patras
  - GSK Investigational Site, Thessaloniki
- Spain (3):
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Omenaca F, Merino JM, Tejedor JC, Constantopoulos A, Papaevangelou V, Kafetzis D, Tsirka A, Athanassiadou F, Anagnostakou M, Francois N, Borys D, Schuerman L. Immunization of preterm infants with 10-valent pneumococcal conjugate vaccine. Pediatrics. 2011 Aug;128(2):e290-8. doi: 10.1542/peds.2010-1184. Epub 2011 Jul 4. PMID 21727108
- [Background] Omeneca F et al. Vaccination of pre-term infants with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHID-CV). Abstract presented at the 27th annual ESPID meeting, Brussels, Belgium, 9-13 June 2009.
- [Background] Omeneca F et al. Immunogenicity and safety of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) following primary and booster vaccination in preterm-born children. Abstract presented at Excellence In Paediatrics. Florence, Italy, 3-6 December 2009.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 107737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107737 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For each subject the study duration was approximately 5 months for the active phase (Month 0 untill one month after last vaccination) and 10 months, including the 5 months extended safety follow-up.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/ exclusion criteria, contraindications/ precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Synflorix™ + Infanrix™ Hexa Group II: Mild preterm infants born after a gestation period of 31-36 weeks (217-258 days)
- Synflorix™ + Infanrix™ Hexa Group III: Infants born after a full-term gestation period of more than 36 weeks (more than 258 days)
Period: Overall Study
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Started | 50 | 87 | 149
Completed | 48 | 83 | 139
Not Completed | 2 | 4 | 10
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 5
Not completed — Withdrawal by Subject | 1 | 3 | 2
Not completed — Migrated/moved from study area | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III | Total
Number analyzed (Participants) | 50 | 87 | 149 | 286
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 11.0 (3.2) | 9.5 (1.45) | 9.3 (1.45) | 9.66 (1.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 40 | 62 | 121
  Male | 31 | 47 | 87 | 165
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Etnicity: White - Caucasian/ European heritage | 36 | 77 | 140 | 253
  Race/Etnicity: African heritage/ African american | 2 | 1 | 4 | 7
  Race/Etnicity: American Indian or Alaskan native | 4 | 6 | 2 | 12
  Race/Etnicity: Asian - south east Asian heritage | 0 | 1 | 0 | 1
  Race/Etnicity: White - Arabic/ north African heritage | 1 | 0 | 2 | 3
  Race/Etnicity: Other (unspecified) | 7 | 2 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Core Fever (Rectal Temperature) Greater Than (>) the Cut-off
Description: Fever was measured as rectal temperature. Assessment of occurrences of fever > 39.0 °C was performed post doses 1, 2 and 3 of Synflorix or Infanrix hexa vaccine.
Time Frame: Within 4 days (Days 0-3) after each vaccine dose, administered according to a 3-dose schedule at 2-4-6 months of age (Month 0-2-4)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with the symptom sheet filled-in.
  The analysis was performed, as planned per protocol, according to 2 groups: Preterm (i.e. very and mild preterm infants "Pooled Group I + II") and Full term group (i.e. "Synflorix™ + Infanrix™ Hexa Group III").
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Group I + II: Pooled group consists of very preterm infants and mild preterm infants (Synflorix™ + Infanrix™ hexa Group I and Synflorix™ + Infanrix™ hexa Group II).
Arm/Group | Synflorix™ + Infanrix™ Hexa Group III | Pooled Group I + II
Number analyzed (Participants) | 146 | 135
Participants
  Fever > 39.0°C, post Dose 1 | 5 | 2
  Fever > 39.0°C, post Dose 2: number analyzed (Participants) | 141 | 133
  Fever > 39.0°C, post Dose 2 | 1 | 1
  Fever > 39.0°C, post Dose 3: number analyzed (Participants) | 138 | 131
  Fever > 39.0°C, post Dose 3 | 3 | 1

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed included pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/ spontaneously painful. Grade 3 swelling/ redness was defined as swelling/ redness greater than (>) 30 millimeters (mm). "Any" was defined as incidence of the specified symptom regardless of intensity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group III | Pooled Group I + II
Number analyzed (Participants) | 146 | 135
Participants
  Any pain, Post Dose 1 | 58 | 40
  Grade 3 pain, Post Dose 1 | 6 | 6
  Any redness, Post Dose 1 | 67 | 39
  Grade 3 redness, Post Dose 1 | 0 | 1
  Any swelling, Post Dose 1 | 67 | 30
  Grade 3 swelling, Post Dose 1 | 2 | 1
  Any pain, Post Dose 2: number analyzed (Participants) | 141 | 133
  Any pain, Post Dose 2 | 39 | 39
  Grade 3 pain, Post Dose 2: number analyzed (Participants) | 141 | 133
  Grade 3 pain, Post Dose 2 | 1 | 9
  Any redness, Post Dose 2: number analyzed (Participants) | 141 | 133
  Any redness, Post Dose 2 | 72 | 41
  Grade 3 redness, Post Dose 2: number analyzed (Participants) | 141 | 133
  Grade 3 redness, Post Dose 2 | 7 | 0
  Any swelling, Post Dose 2: number analyzed (Participants) | 141 | 133
  Any swelling, Post Dose 2 | 60 | 30
  Grade 3 swelling, Post Dose 2: number analyzed (Participants) | 141 | 133
  Grade 3 swelling, Post Dose 2 | 4 | 0
  Any pain, Post Dose 3: number analyzed (Participants) | 138 | 131
  Any pain, Post Dose 3 | 42 | 30
  Grade 3 pain, Post Dose 3: number analyzed (Participants) | 138 | 131
  Grade 3 pain, Post Dose 3 | 6 | 3
  Any redness, Post Dose 3: number analyzed (Participants) | 138 | 131
  Any redness, Post Dose 3 | 66 | 33
  Grade 3 redness, Post Dose 3: number analyzed (Participants) | 138 | 131
  Grade 3 redness, Post Dose 3 | 9 | 3
  Any swelling, Post Dose 3: number analyzed (Participants) | 138 | 131
  Any swelling, Post Dose 3 | 58 | 24
  Grade 3 swelling, Post Dose 3: number analyzed (Participants) | 138 | 131
  Grade 3 swelling, Post Dose 3 | 6 | 2

3. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms
Description: Solicited general symptoms assessed included drowsiness, fever (defined as rectal temperature ≥ 38.0°C), irritability, and loss of appetite. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (rectal temperature) above (>) 40.0 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/ preventing normal activity. Grade 3 loss of appetite was defined as the subject not eating at all. "Any" was defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group III | Pooled Group I + II
Number analyzed (Participants) | 146 | 135
Participants
  Any drowsiness, Post Dose 1 | 53 | 44
  Grade 3 drowsiness, Post Dose 1 | 2 | 1
  Any fever(rectally), Post Dose 1 | 38 | 41
  Grade 3 fever(rectally), Post Dose 1 | 1 | 0
  Any irritability, Post Dose 1 | 73 | 53
  Grade 3 irritability, Post Dose 1 | 9 | 6
  Any loss of appetite, Post Dose 1 | 36 | 33
  Grade 3 loss of appetite, Post Dose 1 | 0 | 0
  Any drowsiness, Post Dose 2: number analyzed (Participants) | 141 | 133
  Any drowsiness, Post Dose 2 | 34 | 32
  Grade 3 drowsiness, Post Dose 2: number analyzed (Participants) | 141 | 133
  Grade 3 drowsiness, Post Dose 2 | 0 | 1
  Any fever(rectally), Post Dose 2: number analyzed (Participants) | 141 | 133
  Any fever(rectally), Post Dose 2 | 34 | 40
  Grade 3 fever(rectally), Post Dose 2: number analyzed (Participants) | 141 | 133
  Grade 3 fever(rectally), Post Dose 2 | 0 | 0
  Any irritability, Post Dose 2: number analyzed (Participants) | 141 | 133
  Any irritability, Post Dose 2 | 53 | 51
  Grade 3 irritability, Post Dose 2: number analyzed (Participants) | 141 | 133
  Grade 3 irritability, Post Dose 2 | 2 | 4
  Any loss of appetite, Post Dose 2: number analyzed (Participants) | 141 | 133
  Any loss of appetite, Post Dose 2 | 23 | 35
  Grade 3 loss of appetite, Post Dose 2: number analyzed (Participants) | 141 | 133
  Grade 3 loss of appetite, Post Dose 2 | 0 | 2
  Any drowsiness, Post Dose 3: number analyzed (Participants) | 138 | 131
  Any drowsiness, Post Dose 3 | 22 | 18
  Grade 3 drowsiness, Post Dose 3: number analyzed (Participants) | 138 | 131
  Grade 3 drowsiness, Post Dose 3 | 1 | 4
  Any fever(rectally), Post Dose 3: number analyzed (Participants) | 138 | 131
  Any fever(rectally), Post Dose 3 | 25 | 16
  Grade 3 fever(rectally), Post Dose 3: number analyzed (Participants) | 138 | 131
  Grade 3 fever(rectally), Post Dose 3 | 1 | 0
  Any irritability, Post Dose 3: number analyzed (Participants) | 138 | 131
  Any irritability, Post Dose 3 | 44 | 40
  Grade 3 irritability, Post Dose 3: number analyzed (Participants) | 138 | 131
  Grade 3 irritability, Post Dose 3 | 1 | 3
  Any loss of appetite, Post Dose 3: number analyzed (Participants) | 138 | 131
  Any loss of appetite, Post Dose 3 | 22 | 26
  Grade 3 loss of appetite, Post Dose 3: number analyzed (Participants) | 138 | 131
  Grade 3 loss of appetite, Post Dose 3 | 0 | 1

4. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" was defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Within 31 days (Days 0-30) after each vaccine dose, administered according to a 3-dose schedule at 2-4-6 months of age (Month 0-2-4)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
  The analysis was performed, as planned per protocol, according to 2 groups: Preterm (i.e. very and mild preterm infants "Pooled Group I + II") and Full term group (i.e. "Synflorix™ + Infanrix™ Hexa Group III").
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group III | Pooled Group I + II
Number analyzed (Participants) | 149 | 137
Participants | 58 | 43

5. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed included medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/ incapacity.
Time Frame: Throughout the active phase of the study (from the first vaccine administration (Month 0) up to 1 month after the third vaccine administration (Month5).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group III | Pooled Group I + II
Number analyzed (Participants) | 149 | 137
Participants | 13 | 18

6. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: as for outcome 5
Time Frame: Throughout the entire study period starting from the first vaccine dose administration (Month 0) up to the end of the 6-month safety follow-up (ESFU- Month 10).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group III | Pooled Group I + II
Number analyzed (Participants) | 149 | 137
Participants | 19 | 29

7. Secondary Outcome: Number of Subjects With Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Greater Than or Equal to (≥) the Cut-off
Description: The cut-off for the assay was ≥ 0.20 microgram per mililiter (μg/ mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort of immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 42 | 82 | 132
Participants
  Anti-1: number analyzed (Participants) | 42 | 82 | 130
  Anti-1 | 41 | 82 | 129
  Anti-4: number analyzed (Participants) | 41 | 82 | 130
  Anti-4 | 40 | 81 | 130
  Anti-5: number analyzed (Participants) | 42 | 82 | 129
  Anti-5 | 42 | 82 | 129
  Anti-6B: number analyzed (Participants) | 41 | 82 | 132
  Anti-6B | 38 | 78 | 123
  Anti-7F: number analyzed (Participants) | 41 | 82 | 132
  Anti-7F | 41 | 82 | 131
  Anti-9V: number analyzed (Participants) | 41 | 82 | 132
  Anti-9V | 40 | 82 | 132
  Anti-14: number analyzed (Participants) | 41 | 82 | 132
  Anti-14 | 41 | 82 | 132
  Anti-18C: number analyzed (Participants) | 41 | 81 | 132
  Anti-18C | 41 | 81 | 130
  Anti-19F | 42 | 82 | 132
  Anti-23F: number analyzed (Participants) | 41 | 82 | 132
  Anti-23F | 39 | 79 | 125

8. Secondary Outcome: Number of Subjects With Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F ≥ the Cut-off
Description: The cut-off for the assay was ≥ 0.05 microgram per mililiter (μg/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: The analysis was performed on the ATP cohort of immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 42 | 82 | 132
Participants
  Anti-1: number analyzed (Participants) | 42 | 82 | 130
  Anti-1 | 42 | 82 | 130
  Anti-4: number analyzed (Participants) | 41 | 82 | 130
  Anti-4 | 41 | 82 | 130
  Anti-5: number analyzed (Participants) | 42 | 82 | 129
  Anti-5 | 42 | 82 | 129
  Anti-6B: number analyzed (Participants) | 41 | 82 | 131
  Anti-6B | 40 | 81 | 131
  Anti-7F: number analyzed (Participants) | 41 | 82 | 131
  Anti-7F | 41 | 82 | 131
  Anti-9V: number analyzed (Participants) | 41 | 82 | 132
  Anti-9V | 41 | 82 | 132
  Anti-14: number analyzed (Participants) | 41 | 82 | 132
  Anti-14 | 41 | 82 | 132
  Anti-18C: number analyzed (Participants) | 41 | 81 | 132
  Anti-18C | 41 | 81 | 131
  Anti-19F | 42 | 82 | 132
  Anti-23F: number analyzed (Participants) | 41 | 82 | 131
  Anti-23F | 39 | 81 | 129

9. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: Seropositivity status, defined as anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 42 | 82 | 132
μg/mL
  Anti-1: number analyzed (Participants) | 42 | 82 | 130
  Anti-1 | 0.97 [0.75 to 1.26] | 1.1 [0.93 to 1.3] | 1.35 [1.18 to 1.55]
  Anti-4: number analyzed (Participants) | 41 | 82 | 130
  Anti-4 | 1.53 [1.19 to 1.98] | 1.88 [1.61 to 2.2] | 2.42 [2.13 to 2.74]
  Anti-5: number analyzed (Participants) | 42 | 82 | 129
  Anti-5 | 1.45 [1.13 to 1.86] | 1.93 [1.65 to 2.25] | 2.31 [2 to 2.66]
  Anti-6B: number analyzed (Participants) | 41 | 82 | 131
  Anti-6B | 0.85 [0.61 to 1.19] | 1.11 [0.89 to 1.37] | 1.18 [1 to 1.39]
  Anti-7F: number analyzed (Participants) | 41 | 82 | 131
  Anti-7F | 1.87 [1.47 to 2.39] | 2.37 [2.07 to 2.73] | 2.69 [2.39 to 3.03]
  Anti-9V: number analyzed (Participants) | 41 | 82 | 132
  Anti-9V | 1.43 [1.17 to 1.74] | 1.69 [1.44 to 1.99] | 2.41 [2.13 to 2.73]
  Anti-14: number analyzed (Participants) | 41 | 82 | 132
  Anti-14 | 3.52 [2.81 to 4.42] | 3.28 [2.77 to 3.89] | 3.71 [3.21 to 4.3]
  Anti-18C: number analyzed (Participants) | 41 | 81 | 132
  Anti-18C | 3.28 [2.51 to 4.29] | 4.86 [3.92 to 6.02] | 5.22 [4.27 to 6.38]
  Anti-19F | 3.6 [2.83 to 4.57] | 4.8 [4.15 to 5.55] | 4.56 [3.95 to 5.26]
  Anti-23F: number analyzed (Participants) | 41 | 82 | 131
  Anti-23F | 1.05 [0.74 to 1.49] | 1.33 [1.07 to 1.65] | 1.54 [1.28 to 1.85]

10. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F ≥ the Cut-off
Description: The cut-off for the assay was ≥ 8
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 36 | 74 | 113
Participants
  Opsono-1: number analyzed (Participants) | 34 | 72 | 110
  Opsono-1 | 20 | 49 | 80
  Opsono-4: number analyzed (Participants) | 36 | 73 | 111
  Opsono-4 | 36 | 72 | 110
  Opsono-5: number analyzed (Participants) | 34 | 74 | 109
  Opsono-5 | 29 | 69 | 104
  Opsono-6B: number analyzed (Participants) | 35 | 69 | 104
  Opsono-6B | 30 | 59 | 85
  Opsono-7F | 36 | 74 | 113
  Opsono-9V: number analyzed (Participants) | 36 | 72 | 103
  Opsono-9V | 36 | 72 | 103
  Opsono-14: number analyzed (Participants) | 36 | 73 | 112
  Opsono-14 | 36 | 73 | 110
  Opsono-18C: number analyzed (Participants) | 34 | 68 | 102
  Opsono-18C | 34 | 65 | 99
  Opsono-19F: number analyzed (Participants) | 35 | 74 | 110
  Opsono-19F | 31 | 71 | 105
  Opsono-23F: number analyzed (Participants) | 36 | 72 | 109
  Opsono-23F | 35 | 70 | 109

11. Secondary Outcome: Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: Seropositivity status, defined as Opsonophagocytic activity against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F ≥ 8.
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 36 | 74 | 113
Titers
  Opsono-1: number analyzed (Participants) | 34 | 72 | 110
  Opsono-1 | 23 [13 to 40.6] | 30.3 [20.5 to 44.8] | 46.3 [33.4 to 64.1]
  Opsono-4: number analyzed (Participants) | 36 | 73 | 111
  Opsono-4 | 644.1 [474.6 to 874] | 500.9 [384.5 to 652.5] | 543.5 [450.6 to 655.5]
  Opsono-5: number analyzed (Participants) | 34 | 74 | 109
  Opsono-5 | 45.2 [27.7 to 73.8] | 70.8 [52.3 to 95.7] | 94.8 [75.7 to 118.7]
  Opsono-6B: number analyzed (Participants) | 35 | 69 | 104
  Opsono-6B | 278.3 [125.5 to 617.3] | 305.1 [180.1 to 516.9] | 268.2 [167.5 to 429.4]
  Opsono-7F | 4086.3 [2834.3 to 5891.3] | 3047.3 [2422.2 to 3833.7] | 2395.2 [1973.2 to 2907.5]
  Opsono-9V: number analyzed (Participants) | 36 | 72 | 103
  Opsono-9V | 930.5 [603.1 to 1435.6] | 837.9 [642.7 to 1092.3] | 1144.8 [922.3 to 1421]
  Opsono-14: number analyzed (Participants) | 36 | 73 | 112
  Opsono-14 | 775.4 [539 to 1115.5] | 901.6 [699.8 to 1161.6] | 644.6 [514.9 to 807]
  Opsono-18C: number analyzed (Participants) | 34 | 68 | 102
  Opsono-18C | 262.5 [159.4 to 432.4] | 321.5 [220.9 to 467.7] | 251 [189 to 333.4]
  Opsono-19F: number analyzed (Participants) | 35 | 74 | 110
  Opsono-19F | 104.2 [61.5 to 176.5] | 201.1 [149.7 to 270.1] | 182.7 [139.2 to 239.7]
  Opsono-23F: number analyzed (Participants) | 36 | 72 | 109
  Opsono-23F | 1659.4 [975.1 to 2824] | 1147.2 [843 to 1561.2] | 1558.8 [1302.6 to 1865.3]

12. Secondary Outcome: Number of Subjects With Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A ≥ the Cut-off
Description: The cut-off for the assay was ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 42 | 81 | 131
Participants
  Anti-6A: number analyzed (Participants) | 42 | 81 | 129
  Anti-6A | 32 | 68 | 114
  Anti-19A | 26 | 72 | 120

13. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Seropositivity status was defined as anti-pneumococcal cross-reactive serotypes 6A and 19A antibody concentrations ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 42 | 81 | 131
μg/mL
  Anti-6A: number analyzed (Participants) | 42 | 81 | 129
  Anti-6A | 0.14 [0.09 to 0.2] | 0.21 [0.15 to 0.28] | 0.2 [0.16 to 0.25]
  Anti-19A | 0.08 [0.06 to 0.11] | 0.21 [0.16 to 0.28] | 0.26 [0.21 to 0.32]

14. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes 6A and 19A ≥ the Cut-off
Description: The cut-off for the assay was ≥ 8.
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 33 | 69 | 105
Participants
  Opsono-6A: number analyzed (Participants) | 33 | 66 | 96
  Opsono-6A | 25 | 54 | 58
  Opsono-19A: number analyzed (Participants) | 31 | 69 | 105
  Opsono-19A | 2 | 10 | 17

15. Secondary Outcome: Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Seropositivity status was defined as opsonophagocytic activity against pneumococcal cross-reactive serotypes 6A and 19A ≥ 8.
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 33 | 69 | 105
Titers
  Opsono-6A | 114.5 [52.8 to 248.5] | 157.3 [95.8 to 258.4] | 49.5 [31.8 to 76.9]
  Opsono-19A: number analyzed (Participants) | 31 | 69 | 105
  Opsono-19A | 4.5 [3.8 to 5.4] | 7.1 [4.9 to 10.1] | 7 [5.4 to 9.2]

16. Secondary Outcome: Number of Subjects With Concentrations of Antibodies Against Protein D (Anti-PD) ≥ the Cut-off
Description: The cut-off for the assay was ≥ 100 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 42 | 82 | 130
Participants | 42 | 82 | 130

17. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD)
Description: Seropositivity status was defined as anti-PD antibody concentrations ≥ 100 ELISA units per milliliter ( EL.U/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 42 | 82 | 130
EL.U/mL | 1688.6 [1320.1 to 2159.8] | 1415.4 [1167.1 to 1716.5] | 1496.8 [1283.4 to 1745.8]

18. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti DT) and Anti-tetanus Toxoids (Anti TT) Antibody Concentrations ≥ the Cut-off
Description: The cut-off for the assay was ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 18 | 41 | 61
Participants
  Anti-diphtheria | 18 | 41 | 61
  Anti-tetanus | 18 | 41 | 61

19. Secondary Outcome: Antibody Concentrations for Anti-diphtheria and Tetanus Toxoids ≥ the Cut-off
Description: Seroprotection status was defined as anti-diphtheria toxoid or anti-tetanus toxoid antibody concentrations ≥ 0.1 IU/mL
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 18 | 41 | 61
IU/mL
  Anti-diphtheria | 2.495 [1.664 to 3.741] | 3.23 [2.628 to 3.969] | 3.077 [2.481 to 3.817]
  Anti-tetanus | 7.745 [6.284 to 9.545] | 8.617 [7.216 to 10.29] | 7.695 [6.838 to 8.66]

20. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration ≥ the Cut-off
Description: The cut-off for the assay was ≥ 0.15 microgram per milliliter (μg/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 18 | 41 | 63
Participants | 18 | 41 | 63

21. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration ≥ the Cut-off
Description: The cut-off for the assay was ≥ 1.0 microgram per milliliter (μg/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 18 | 41 | 63
Participants | 16 | 38 | 60

22. Secondary Outcome: Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibody Concentrations ≥ th Cut-off
Description: Seroprotection status was defined as anti-PRP antibody concentrations ≥ 0.15 μg/mL and ≥ 1.0 μg/mL
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 18 | 41 | 63
μg/mL | 4.031 [2.261 to 7.184] | 5.804 [4.12 to 8.178] | 7.952 [5.839 to 10.831]

23. Secondary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations ≥ the Cut-off
Description: The cut-off for the assay was ≥ 5 ELISA unit per milliliter (EL.U/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 18 | 41 | 61
Participants
  Anti-PT | 18 | 41 | 61
  Anti-FHA | 18 | 41 | 61
  Anti-PRN: number analyzed (Participants) | 17 | 40 | 60
  Anti-PRN | 17 | 40 | 60

24. Secondary Outcome: Antibody Concentration for Anti-pertussis Toxoid (Anti-PT) , Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: Seropositivity status was defined as anti-PT, anti-FHA, anti-PRN antibody concentrations ≥ 5 EL.U/mL.
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 18 | 41 | 61
EL.U/mL
  Anti-PT | 41.9 [27.6 to 63.7] | 37.9 [30.7 to 46.7] | 47.3 [40.2 to 55.7]
  Anti-FHA | 188.6 [133.4 to 266.6] | 169 [139.6 to 204.7] | 163.1 [138.3 to 192.3]
  Anti-PRN: number analyzed (Participants) | 17 | 40 | 60
  Anti-PRN | 127.6 [81.5 to 199.6] | 109.1 [85.7 to 139] | 119.1 [101.1 to 140.4]

25. Secondary Outcome: Number of Subjects With Anti-Hepatitis B Surface Antigen (HBs) Antibody Concentrations ≥ the Cut-off.
Description: The cut-off for the assay was ≥ 10 milli-international units per milliliter (mIU/mL).
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 8 | 26 | 12
Participants | 8 | 26 | 12

26. Secondary Outcome: Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations
Description: Seroprotection status was defined as Anti-HBs antibody concentrations ≥ 10 mIU/mL
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 8 | 26 | 12
mIU/mL | 431.9 [240.7 to 775.2] | 356 [221.1 to 573.4] | 462.9 [221.1 to 969.1]

27. Secondary Outcome: Number of Subjects With Anti-polio Type 1, 2 and 3 Antibody Titres
Description: The cut-off for the assay was ≥ 8.
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 12 | 22 | 29
Participants
  Anti-Polio 1 | 12 | 22 | 29
  Anti-Polio 2 | 12 | 22 | 29
  Anti-Polio 3: number analyzed (Participants) | 11 | 21 | 29
  Anti-Polio 3 | 10 | 21 | 29

28. Secondary Outcome: Antibody Titers for Polio Type 1, 2 and 3 ≥ the Cut-off
Description: Seroprotection status was defined as Anti-polio type 1, Anti-polio type 2 and Anti-polio type 3 antibody titers ≥ 8.
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 12 | 22 | 29
Titers
  Anti-Polio 1 | 271.3 [132.9 to 554] | 189.5 [109.9 to 326.8] | 230.1 [166 to 319]
  Anti-Polio 2 | 341.7 [214 to 545.6] | 319 [172.5 to 589.8] | 194.4 [121.7 to 310.7]
  Anti-Polio 3 | 248.4 [67.9 to 908.7] | 344.7 [192.2 to 618.3] | 384.8 [245.3 to 603.6]

29. Secondary Outcome: Number of Subjects With Vaccine Response to Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: Vaccine response to PT, FHA and PRN was defined as appearance of antibodies in subjects who are initially seronegative (S-), or at least maintenance of pre-vaccination antibody concentrations in those who are initially seropositive (S+). For the SYNFLORIX™ + INFANRIX™ HEXA GROUP I, no subjects presented initial seropositivity for PT and PRN antigens.
Time Frame: One month after the 3rd vaccine dose (Month 5)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
Number analyzed (Participants) | 18 | 34 | 45
Participants
  Anti-PT, S- | 18 | 27 | 45
  Anti-PT, S+: number analyzed (Participants) | 0 | 10 | 13
  Anti-PT, S+ | 0 | 8 | 12
  Anti-FHA, S-: number analyzed (Participants) | 15 | 22 | 18
  Anti-FHA, S- | 15 | 22 | 18
  Anti-FHA, S+: number analyzed (Participants) | 3 | 17 | 41
  Anti-FHA, S+ | 3 | 17 | 41
  Anti-PRN, S-: number analyzed (Participants) | 17 | 34 | 45
  Anti-PRN, S- | 17 | 34 | 45
  Anti-PRN, S+: number analyzed (Participants) | 0 | 4 | 12
  Anti-PRN, S+ | 0 | 4 | 12

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day post vaccination; Unsolicited AEs: during the 31-day post vaccination; SAEs: during the whole study period (Month 0 - Month 10, including the 5 months extended safety follow-up).
Arm/Group | Synflorix™ + Infanrix™ Hexa Group I | Synflorix™ + Infanrix™ Hexa Group II | Synflorix™ + Infanrix™ Hexa Group III
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/87 | 0/149
Serious Adverse Events (participants affected / at risk) | 17/50 | 11/87 | 19/149
Other Adverse Events (participants affected / at risk) | 42/50 | 76/87 | 136/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix™ + Infanrix™ Hexa Group I (N=50) | Synflorix™ + Infanrix™ Hexa Group II (N=87) | Synflorix™ + Infanrix™ Hexa Group III (N=149)
Thrombocythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subdural hygroma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Breath holding (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix™ + Infanrix™ Hexa Group I (N=50) | Synflorix™ + Infanrix™ Hexa Group II (N=87) | Synflorix™ + Infanrix™ Hexa Group III (N=149)
Decreased appetite (Metabolism and nutrition disorders) | 19 (30) | 46 (64) | 51 (81)
Erythema (Skin and subcutaneous tissue disorders) | 24 (32) | 49 (81) | 102 (205)
Injection site nodule (General disorders) | 0 (0) | 4 (4) | 10 (14)
Irritability (Psychiatric disorders) | 22 (38) | 53 (106) | 100 (171)
Pain (General disorders) | 24 (34) | 41 (75) | 84 (139)
Pyrexia (General disorders) | 22 (29) | 45 (70) | 71 (106)
Somnolence (Nervous system disorders) | 20 (30) | 44 (64) | 65 (109)
Swelling (General disorders) | 20 (27) | 35 (57) | 98 (185)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 9 (9) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.